CLINICAL TRIAL: NCT00973674
Title: A Phase II Trial to Evaluate the Effects of A Single Dose of Intravenous Premarin for the Treatment of Severe Traumatic Brain Injury
Brief Title: Resuscitative Endocrinology:Single-dose Clinical Uses for Estrogen-Traumatic Brain Injury
Acronym: RESCUE-TBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Washington (Other); Resuscitation Outcomes Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESCUE-TBI
Record Dates: First submitted 2009-07-14; First posted 2009-09-09 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Estrogens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Premarin IV (Experimental): Patients randomized to receive a single dose of 0.5 mg/kg Premarin® IV
  Interventions: Drug: Premarin IV
- Placebo (Placebo Comparator): Patients randomized to receive a single dose of placebo IV. Due of the faint yellow color of the reconstituted Premarin®, the placebo dose will be prepared with 0.14 ml of Vial 1 of Infuvite Adult Multivitamin and 14 ml of sterile water to generate a similar color and volume. This aliquot will be used only for those study patients who are randomized to the placebo arm. The placebo volume will be approximately equal to the volume which the patient would have received had the patient been randomized to the Premarin arm Considering the small amount of IV multivitamin needed for fluid tinting, it is not expected that the IV multivitamin will have any effect on patients with traumatic brain injury.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Premarin IV — One time dose of Premarin IV
  Other Names: IV Estrogen
  Arms: Premarin IV
Drug: Placebo — One time dose of Placebo
  Other Names: Infivite Multivitamin
  Arms: Placebo

SUMMARY:
Each year in the United States alone, a third of a million persons are hospitalized for traumatic brain injury (TBI), of whom approximately 1/4 die. Most are less than 30 years of age. Not only are the health care costs staggering for both initial care and rehabilitation, but the societal loss in terms of economic impact reaches into the billions of dollars annually in the U.S. alone. Despite advances in neurosurgical interventions and intensive care management, many survivors do not fully recover. A significant cause of this mortality and morbidity is thought due to potentially preventable secondary injury, namely oxidant injury, inflammation, and apoptosis in the penumbra (the area of brain surrounding the primary lesion, which is at-risk, but potentially salvageable), beginning in the first few hours after the severe traumatic event.

Despite the current bleak outlook for many of these patients, a series of animal investigations have uncovered a promising solution to the problem of the secondary injury seen in severe TBI and other similar processes, namely the early administration of estrogen, a strong anti-oxidant, anti-inflammatory and anti-apoptotic compound. Based on these encouraging results from animal studies, the investigators hypothesize that early administration of IV Premarin® in patients with severe TBI will safely reduce secondary brain injury, improve neurological outcomes, and improve survival.

DETAILED DESCRIPTION:
Early estrogen treatment has been tested in a myriad of animal models of resuscitation ranging from TBI and stroke to spinal cord injury, trauma-related hemorrhage, and sepsis. In these scenarios, studies using old and young, male and female animals found estrogen to be a strikingly effective therapy. Importantly, various animal studies examining brain injury sizes via radiological imaging and sophisticated immunofluorescent techniques have revealed significant protective effects of IV estrogen given post-injury, noting decreases in injury size of up to 65% in those receiving estrogen compared with those not receiving it. Furthermore, this beneficial effect is seen in all body tissues in both males and females. Only one identified TBI study to date did not show similar efficacy. A rodent model of TBI found that all females, in all three groups (those receiving no treatment, placebo, and estrogen) inexplicably died.

Mechanisms of Estrogen's Neuroprotection The use of estrogen as an acute resuscitation drug for severe brain injury has been extensively investigated in animal models. The mechanisms of estrogen's protective effects are numerous, including prevention of propogation of oxidant injury, anti-inflammatory properties in all major organs in the body, and mitochondria stabilization.

Importantly, the following studies find that estrogen exerts significant neuroprotective effects aimed at many of the mechanisms implicated in devastating secondary brain injury in TBI, including:

Brain Ischemia and Reperfusion Intracerebral Hemorrhage (a frequent component of traumatic brain injury) Impaired Cerebral Blood Flow Cerebral Vasospasm Cerebral Metabolic Dysfunction, including mitochondrial dysfunction with reduction of ATP production Cerebral Excitotoxicity and Blood Brain Barrier Preservation Cerebral Oxidant Injury Cerebral Edema Cerebral Inflammation Apoptosis

The protective effects of estrogen may initially appear counterintuitive in light of the recent WHI and HERS trials which studied long-term, oral, low-dose administration of estrogen in older, significantly-post menopausal women. In contrast, the proposed study utilizes a one-time resuscitative dose of IV estrogen administered rapidly following the injury. From a safety standpoint, there are a hundred-million women years of safety data for estrogen's clinical use, and safe use has been documented in men with prostate cancer, uremic bleeding, liver transplantation, and spine surgery. Any safety concerns, such as clotting effects found with long-tem, orally administered estrogen would not be expected when administered one time through an IV dose. Estrogen, when administered IV, avoids the first pass effect in the liver, and does not trigger the ER-α mediated pro-thrombotic effects seen with oral administration. Therefore, it is felt that this acute, IV single-dose administration of estrogen will convey the protective benefits seen in animal studies without side effects implicated with long-term oral use in humans.

Finally, estrogen is not the only sex steroid implicated in resuscitation. While estrogen has been the most frequently studied sex steroid in animal resuscitation models, progesterone too is thought to have potential neuroprotective effects. There is a recently published clinical pilot trial of IV progesterone as an acute resuscitative therapy for TBI patients, which indicates potentially promising clinical results without negative safety findings, thereby also poising this sex steroid for future multi-center trials.

In summary, we believe that there are compelling reasons to evaluate estrogen as an acute intervention in patients with traumatic brain injury given the benefit demonstrated in animal studies of brain injury, and safety data in humans prescribed estrogen for other indications. But we are aware that there are no published data related to use of a single dose of IV estrogen in injured patients in the acute setting. Therefore we have conceptualized our trial with frequent evaluation of patient safety through an organized Data Safety Monitoring Committee.

Potential participants include patients between the ages of 18 and 55 years who are admitted to Parkland Memorial Hospital or Baylor University Medical Center with a presumed diagnosis of severe traumatic brain injury. This young population was chosen for several reasons:

1. This population represents the most frequent patient with TBI (young).
2. This population filters out confounders such as chronic, age-related illnesses. Upon admission to the Emergency Department and evaluation of the patient in light of study criteria, qualified participants will be randomized to receive a single dose of 0.5 mg/kg Premarin® IV or placebo. One 7cc tube of blood and available urine will be drawn for baseline values prior to study drug administration. Those patients who require the placement of a ventriculostomy by a neurosurgeon for therapeutic treatment will also have one 7cc test tube of blood and available urine from the foley catheter drawn at the time the ventriculostomy is placed. Upon placement of the ventriculostomy, cerebral spinal fluid that would otherwise be discarded will be collected. These fluids will be centrifuged and frozen within one hour of collection, and the blood, CSF and urine analyzed in batches for markers of injury and repair. These samples will then be serially collected on an every four hour schedule over the first 24 hours, then every 8 hours for the following 4 days. CSF collection will end early if the ventriculostomy is removed for clinical reasons. Clinically-relevant patient progress (such as vital signs, Glasgow Coma Scale (GCS), partial pressure of carbon dioxide in the arterial blood (PaCO2), intracranial pressure (ICP), and temperature), clinically required interventions, neuro-imaging results, and demographics will be monitored and tracked.

For assessing length of time in coma and orientation, we will administer the Galveston Orientation and Amnesia Test (GOAT) daily until the patient successfully completes the test, for up to 2 months.

Longer-term neurological outcomes will be measured at discharge, 28 days, 3 and 6 months post-injury utilizing the Disability Rating Scale, Glasgow Outcome Score-Extended (GOSE), and Functional Status Examination. These outcomes measures will be collected by the research staff via telephone interviews if the patient has been discharged. The Disability Rating Scale (DRS), Glasgow Outcome Scale-Extended GOSE, and Functional Status Examination are well validated in the literature for follow-up in patients with TBI. These tests can be easily administered over the phone to either the patient or the caregiver.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected blunt head injury
2. Estimated age of 18 - 50 years
3. Estimated time to study drug administration < 2 hours post-trauma
4. Glasgow Come Scale (GCS) score of between 3 and 8 prior to intubation and/or sedation, due to difficulty of patient's cooperation in assessment after these interventions.
5. Systolic blood pressure > 90 mm Hg
6. Receiving medical treatment in the Emergency Department (ED) of Parkland Hospital, or Baylor University Medical Center Emergency Department, Level I Trauma Centers in Dallas,Texas

Exclusion Criteria:

1. Legal Do Not Resuscitate (DNR) orders in place prior to randomization.
2. Known incarcerated individuals
3. Status epilepticus prior to study drug administration
4. Penetrating head trauma
5. Estimated time to study drug administration > 2 hours post-trauma
6. Injury time unknown
7. Cardiopulmonary Resuscitation (CPR) prior to study drug administration
8. Severe hypothermia (suspected T <28C)
9. Drowning or asphyxia due to hanging
10. Burns TBSA > 20% in adults
11. Known inclusion in another interventional trial related to this traumatic event prior to randomization
12. Systolic blood pressure < or = 90 mm Hg
13. Known indication for IV estrogen
14. Known contraindication for estrogen (male sex is NOT a contraindication)
15. Sustained pulse oximeter < 90
16. Recognized spinal cord injury prior to study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane G Wigginton, MD, Principal Investigator — UT Southwestern Medical Center Dallas; Schmickers Rob, Study Chair — University of Washington
Locations (2):
- United States (2):
  - Parkland Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical sites enrolled men and women age 18 to 55 who experienced severe traumatic brain injury in the EMS setting between September 2009 and January 2012.
Groups:
- Placebo: Patients randomized to receive a single dose of placebo IV. Due to the faint yellow color of the reconstituted Premarin®, the placebo dose will be prepared with 0.14 ml of Vial 1 of Infuvite Adult Multivitamin and 14 ml of sterile water to generate a similar color and volume. This aliquot will be used only for those study patients who are randomized to the placebo arm. The placebo volume will be approximately equal to the volume which the patient would have received had the patient been randomized to the Premarin arm Considering the small amount of IV multivitamin needed for fluid tinting, it is not expected that the IV multivitamin will have any effect on patients with traumatic brain injury.
  Placebo: One time dose of Placebo
Period: Overall Study
Arm/Group | Premarin IV | Placebo
Started | 24 | 26
Completed | 22 | 26
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Premarin IV | Placebo | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Continuous [Mean (Full Range); unit: years] | 31.9 [17 to 52] | 34.3 [16 to 65] | 33.3 [16 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percent Passing the Galveston Orientation Amnesia Test (GOAT) Within 28 Days Post Injury
Description: The GOAT is a measure of early cognitive recovery following a severe traumatic injury. The score is determined after examination by health professionals with respect to orientation to person, place and time. On a scale 0 to 100, 76-100 represents normal recovery. The trial measures the percentage of patients who pass the Galveston Orientation Amnesia Test (GOAT) within 28 days post injury.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 22 | 26
Participants | 12 | 14
Statistical Analysis 1: Comparison: Premarin IV vs Placebo; Test type: Superiority or Other; p = 0.99, Barnard's unconditional Exact Test

2. Secondary Outcome: 28-day Mortality
Description: Mortality is defined as the number of patients who died prior to 28 days post injury. Patients who are still in the hospital 28-days post injury are considered alive. The trial examines the rate of enrolled patients on each arm who died prior to 28 days post injury.
Time Frame: 28 Days
Measure: Number; unit: participants
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 22 | 26
participants | 7 | 2
Statistical Analysis 1: Comparison: Premarin IV vs Placebo; Test type: Superiority or Other; p = .033, Log Rank; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [0.74 to 3.77]

3. Secondary Outcome: 6-month Glasgow Outcomes Scale- Extended (GOSE) Score
Description: The GOSE is a scale for functional outcome following a severe traumatic injury. The GOSE is an ordinal variable with the following categories: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery. The GOSE score is determined by a structured interview with questions surrounding consciousness, independence inside and outside the home, social and leisure activities and return to normal life among others. A higher score is considered to be a better result. A lower score indicates a worse result. The scale is 1-8, level 1 minimum score, level 8 maximum score.
Time Frame: Up to 6 months post-injury
Population: The study specifically measures long-term GOSE, defined as post 6 months. Six month follow-up were not available for all patients and thus the lower sample size. As a secondary measure, missing values were not imputed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 18 | 22
units on a scale | 4.00 (2.85) | 4.82 (2.58)
Statistical Analysis 1: Comparison: Premarin IV vs Placebo; Test type: Superiority or Other; p = .35, t-test, 2 sided

4. Secondary Outcome: Acute Respiratory Distress Syndrome (ARDS) Free Survival
Description: ARDS is a life-threatening condition characterized by inflammation of the lungs. The trial measures the number of days alive and without ARDS within 28 days post injury. Patients who die within 28 days are given value of 0, similarly, patients who live 28 days but have ARDS for all 28 days. A higher score indicates better prognosis.
Time Frame: Days 0-28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Premarin IV | Placebo
Number analyzed (Participants) | 22 | 26
days | 18.9 (13.2) | 24.1 (8.7)

ADVERSE EVENTS:
Arm/Group | Premarin IV | Placebo
Serious Adverse Events (participants affected / at risk) | 8/22 | 13/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premarin IV (N=22) | Placebo (N=26)
Pneumonia (Infections and infestations) | 4 (4) | 9 (9)
Bloodstream infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Line infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolus (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes